CLINICAL TRIAL: NCT01568229
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Add-on AMG 747 on Schizophrenia Negative Symptoms
Brief Title: 20110165: Study to Evaluate the Effect of AMG 747 on Schizophrenia Negative Symptoms (Study 165)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxic Epidermal Necrolysis
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110165; 2011-004845-42 (EudraCT Number)
Record Dates: First submitted 2012-02-28; First posted 2012-04-02 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — (R)-2-(4-(phenyl(3-(trifluoromethyl)phenyl)methyl)piperazin-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMG 747 - Dose 1 (Experimental)
  Interventions: Drug: AMG 747
- AMG 747 - Dose 2 (Experimental)
  Interventions: Drug: AMG 747
- AMG 747 - Dose 3 (Experimental)
  Interventions: Drug: AMG 747
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 747 — Three dose levels once-daily oral administration
  Arms: AMG 747 - Dose 1; AMG 747 - Dose 2; AMG 747 - Dose 3
Drug: Placebo — Once-daily oral administration
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the effect of AMG 747 on negative symptoms of schizophrenia in patients who are stable on current antipsychotic treatment. After a run-in period on their current antipsychotic treatment, patients will be randomized to one of the four treatment arms as add-on therapy for a treatment duration of up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) schizophrenia
* Total score on the PANSS Marder Negative Symptom Factor Scale (NSFS) ≥ 20
* Total score on the PANSS Marder Positive Symptom Factor Scale (PSFS) ≤ 30
* Receiving stable antipsychotic therapy for at least 8 weeks prior to screening
* Receiving a stable dose of other psychotropic agents for at least 8 weeks prior to screening
* Subject has had a stable residence or living arrangement for at least 8 weeks prior to screening and the residence or living arrangement is not anticipated to change for the duration of the study
* The subject or subject's legally acceptable representative has provided informed consent.

Exclusion Criteria:

* Current schizoaffective or bipolar disorder, panic disorder, obsessive compulsive disorder, evidence of mental retardation by history or clinical examination or known premorbid IQ ≤ 70
* Clinically significant suicidal ideation or suicide attempts, assaultive behavior or marked changes in mood within the 8 weeks prior to screening, or currently endorsing suicidal ideation in clinical exam
* Substance abuse (with the exception of nicotine or caffeine abuse) within the 8 weeks prior to screening, or during screening
* Substance dependence (with the exception of nicotine or caffeine dependence) within the 6 months prior to screening, or during screening
* Planning to initiate a smoking cessation therapy or otherwise substantially modify nicotine use during the study
* Positive urine drug test for substances of abuse (with the exception of positive screens for prescribed agents such as benzodiazepines).
* Other criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 in negative symptoms, as measured by the NSA-16 total score | 12 Weeks
  NSA-16 = 16-item Negative Symptom Assessment Scale, an efficacy scale used for the primary endpoint

SECONDARY OUTCOMES:
Response defined as a ≥ 20% decrease in the NSA-16 total score at week 12 | 12 Weeks
  NSA-16 = 16-item Negative Symptom Assessment Scale
Change from baseline to week 12 on the PANSS total score and Marder factor scores | 12 weeks
  Positive and Negative Syndrome Scale (PANSS)
Change from baseline to week 12 on the CGI-S | 12 weeks
  Clinical Global Impression Severity Scale (CGI-S)
CGI-I scores at week 12 | 12 weeks
  Clinical Global Impression Improvement (CGI-I)
Change on cognition battery | 12 weeks
Change in personal and social functioning | 12 weeks
Change on patient reported outcomes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (17):
  - Research Site, Little Rock, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Oakland, California
  - Research Site, Orange, California
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Rockville, Maryland
  - Research Site, Flowood, Mississippi
  - Research Site, Princeton, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Scranton, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
- Czechia (5):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Přerov
  - Research Site, Strakonice
- France (4):
  - Research Site, Créteil
  - Research Site, Dôle
  - Research Site, Montauban
  - Research Site, Nîmes
- Malaysia (2):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Ipoh, Perak
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Chełmno
  - Research Site, Katowice
  - Research Site, Skorzewo
  - Research Site, Torun
  - Research Site, Żuromin
- United Kingdom (6):
  - Research Site, Barnet
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Norwich
  - Research Site, Sheffield
  - Research Site, Warrington

REFERENCES:
- [Derived] Dunayevich E, Buchanan RW, Chen CY, Yang J, Nilsen J, Dietrich JM, Sun H, Marder S. Efficacy and safety of the glycine transporter type-1 inhibitor AMG 747 for the treatment of negative symptoms associated with schizophrenia. Schizophr Res. 2017 Apr;182:90-97. doi: 10.1016/j.schres.2016.10.027. Epub 2016 Oct 24. PMID 27789188
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com